CLINICAL TRIAL: NCT04237714
Title: Cultural Adaptation of the Smile is Fun Program for the Treatment of Depression in the Ecuadorian Public Health Care System: A Study Protocol for a Randomized Controlled Trial
Brief Title: Internet-based Intervention Culturally Adapted for Treatment of Depression in the Ecuadorian Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00016-UV-E-2019
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Depression
Keywords: Cultural adaptation; Internet-based intervention; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IBI-based automated support (Experimental): Internet-based intervention with automated support by the system. It consistes in phone text messages twice a week for users. The content of the messages focuses on motivating and reminding users to complete the activities proposed in the program and reviewing the treatment contents. Additionally an automatic email is send if participants have not access the program for a week. The program also provides continuous feedback to users through transversal tools.
  Interventions: Behavioral: Smiling is fun
- IBI-plus human support (Experimental): In this condition, the participants receive automated support explained above and additionally human support for a maximum of 5 minutes that consist in a weekly phone call provided by a psychologist. The content of phone calls is related with resolve questions or doubts about the use and clinical content of the IBI and also motivating and reminding the importance to complete activities in the program.
  Interventions: Behavioral: Smiling is fun
- Control group (No Intervention): Waiting list control group.

INTERVENTIONS:
Behavioral: Smiling is fun — Smile is Fun is a self-applied program that combines elements of prevention and psychological treatment for emotional disorders. It is delivered via the Internet and it is based on CBT technics. The program consists of 8 therapeutic modules and includes 3 transversal tools (activity report, calendar, how am I?) to provide feedback and accompany patients during the intervention. The program requires 8 to 10 weeks to complete in its entirety.
  The intervention, initially developed in Spain, will be adapted to the Ecuadorian culture including elements of the local population, such as, dialect, personal stories, examples and activities. The Ecuadorian version will be evaluate by health professional and users of public health system of Ecuador.
  Arms: IBI-based automated support; IBI-plus human support

SUMMARY:
Internet-Based Interventions are increasingly relevant as an alternative for reducing the gap in treatment of metal disorders such as depression, especially in resource-limited regions.

In this study the investigators will try to evaluate the effectiveness of an Internet-Based Intervention culturally adapted to the Ecuadorian population for treatment of depression.

DETAILED DESCRIPTION:
Our participants will be randomized to one of the following three conditions: 1) Internet-Based intervention (IBI) with automated support (e.g. e-mails or text messages), 2) IBI plus human support by phone calls (automated + human support), 3) Waiting list control group .

The corresponding evaluations of the outcomes will be carried out at different moments of the process: baseline, three, six and twelve months.

This study will use the Smile is Fun program for the treatment of depression previously adapted to the Ecuadorian context.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and read Spanish and access to Internet and having an email address
* Access to a computer or smart phone with internet at home
* Criteria for diagnosis of depression disorder according to the MINI interview and score between 5 to 9 (mild) 10 to 14 (moderate) and 15 to 19 (Moderate/severe) on PHQ-9

Exclusion Criteria:

* Scores 20-27 (severe depression) on PHQ-9
* Suicidal risk
* Severe psychiatric disorders (schizophrenia, substance dependence, bipolar disorder, psychotic illness)
* Receiving psychological treatment for depression at the time of recruitment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in depression symptoms. Beck Depression Inventory- II (BDI-II) | Baseline (week 0), 3, 6 and 12 months.
  It is a 21 item self-report that measure the presence of depressive symptoms in the past two weeks. Spanish version by Sanz et al., 2003.
Change in depression symptoms. Patient Health Questionnaire (PHQ-9) | Baseline (week 0), 3, 6 and 12 months.
  The questionnaire is composed of 9 items, it can be used as a screening test or as an evaluation instrument for depressive disorder. Spanish version by Diez-Quevedo et al., 2001.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder Scale (GAD-7) | Baseline (week 0), 3, 6 and 12 months.
  It is a 7-item scale designed for symptom detection and severity analysis of generalized anxiety disorder. Spanish version by Muñoz-Navarro et al., 2017.
Positive and Negative Affect Schedule (PANAS) | Baseline (week 0), post-module (weekly for 8 weeks), 3, 6 and 12 months.
  This scale consists of 2 subscales, each with 10 items that value positive and negative affects. Spanish version by Lopez-Gomez, Hervas, & Vazquez, 2015.
Overall Anxiety Severity and Impairment Scale (OASIS) | post-module (weekly for 8 weeks)
  This scale has five items related with: the frequency of symptoms of anxiety, their intensity, their interference with the person's work or school life, and their interference with social life. All items are rated on a 5-point Likert scale ranging from 0 (I didn't feel anxious) to 4 (Constant anxiety). Spanish version by Osma, J et al. 2019
Overall Depression Severity and Impairment Scale ODSIS | post-module (weekly for 8 weeks)
  The ODSIS includes five items related with: the frequency of symptoms of depression, their intensity, their interference with the person's work or school life, and their interference with social life. All items are rated on a 5-point Likert scale ranging from 0 (I didn't feel depression) to 4 (Constant depression).
Assessment of Quality of life (AQoL-6D) | Baseline (week 0), 3, 6 and 12 months
  It is a 20-item questionnaire that measures the following dimensions of the patient's health status: illness, independence to live, social relationships, physical and psychological well-being.
Trimbos/iMTA Questionnaire on costs on Psychiatric Illnesses (TIC-P) | Baseline (week 0), 3, 6 and 12 months.
  Questionnaire used to collect information on health services and medication received during the last months, as well as, information on productivity loss in paid and unpaid work depending on the illness.
Client Satisfaction Questionnaire (CSQ-8) | 3 months
  This is a 8-item questionnaire that measures the perception of the attention received. Spanish version by Echeburúa & Corral, 1998
Attitudes Towards Psychological Interventions (APOI) | Baseline (week 0)
  The questionnaire measures expectations towards online psychological interventions. Its 16 items measure: a) skepticism and risk perception, b) confidence in effectiveness, c) risks of technology and d) anonymous benefits.
Credibility and Expectancy Questionnaire (CEQ) | Baseline (week 0)
  This scale is a self-administered 6-item assessment instrument created to measure the belief that the treatment works and the expectations that the treatment will improve.
Semi-structured qualitative interview | post-treatment (8 weeks)
  An Ad-hoc instrument with open questions created to investigate the reasons for abandoning treatment.
Working Alliance Inventory for Online Intervention-Short Form (WAI-TECH- SF) | Baseline (week 0)
  It is a 12-item self-report adapted of the WAI-SF (Hatcher and Gillaspy, 2006). This questionnaire aimed at assessing the working alliance with the online intervention.
System Usability Scale (SUS) | 3 months
  The SUS is a 10-item self-report scale from 0 ("strongly disagree") to 4 ("strongly agree") that measures the usability of a service or product and the acceptance of technology by people who use it.
Semi-structured qualitative interview | 3 months
  A 11-item qualitative interview will be developed. It consists of 6 items rated on a scale from 1 ("very little") to 5 ("very much") and 4 dichotomous questions ("yes" or "no") to assess participants' opinions about the program and the support received.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Baños, PhD, Study Director — University of Valencia
Locations (1):
- Carlos Quiñonez Freire, Santo Domingo, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson G, Carlbring P, Titov N, Lindefors N. Internet Interventions for Adults with Anxiety and Mood Disorders: A Narrative Umbrella Review of Recent Meta-Analyses. Can J Psychiatry. 2019 Jul;64(7):465-470. doi: 10.1177/0706743719839381. Epub 2019 May 16. PMID 31096757
- [Background] Andersson G, Cuijpers P, Carlbring P, Riper H, Hedman E. Guided Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: a systematic review and meta-analysis. World Psychiatry. 2014 Oct;13(3):288-95. doi: 10.1002/wps.20151. PMID 25273302
- [Background] Berger T, Hammerli K, Gubser N, Andersson G, Caspar F. Internet-based treatment of depression: a randomized controlled trial comparing guided with unguided self-help. Cogn Behav Ther. 2011;40(4):251-66. doi: 10.1080/16506073.2011.616531. PMID 22060248
- [Background] Cuijpers P, van Straten A, Andersson G, van Oppen P. Psychotherapy for depression in adults: a meta-analysis of comparative outcome studies. J Consult Clin Psychol. 2008 Dec;76(6):909-22. doi: 10.1037/a0013075. PMID 19045960
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Espinosa HD, Carrasco A, Moessner M, Caceres C, Gloger S, Rojas G, Perez JC, Vanegas J, Bauer S, Krause M. Acceptability Study of "Ascenso": An Online Program for Monitoring and Supporting Patients with Depression in Chile. Telemed J E Health. 2016 Jul;22(7):577-83. doi: 10.1089/tmj.2015.0124. Epub 2016 Jan 7. PMID 26741190
- [Background] Hadjistavropoulos HD, Nugent MM, Alberts NM, Staples L, Dear BF, Titov N. Transdiagnostic Internet-delivered cognitive behaviour therapy in Canada: An open trial comparing results of a specialized online clinic and nonspecialized community clinics. J Anxiety Disord. 2016 Aug;42:19-29. doi: 10.1016/j.janxdis.2016.05.006. Epub 2016 May 13. PMID 27244278
- [Background] Harper Shehadeh M, Heim E, Chowdhary N, Maercker A, Albanese E. Cultural Adaptation of Minimally Guided Interventions for Common Mental Disorders: A Systematic Review and Meta-Analysis. JMIR Ment Health. 2016 Sep 26;3(3):e44. doi: 10.2196/mental.5776. PMID 27670598
- [Background] Bouwmans C, De Jong K, Timman R, Zijlstra-Vlasveld M, Van der Feltz-Cornelis C, Tan Swan S, Hakkaart-van Roijen L. Feasibility, reliability and validity of a questionnaire on healthcare consumption and productivity loss in patients with a psychiatric disorder (TiC-P). BMC Health Serv Res. 2013 Jun 15;13:217. doi: 10.1186/1472-6963-13-217. PMID 23768141
- [Background] Hawthorne G, Richardson J, Osborne R. The Assessment of Quality of Life (AQoL) instrument: a psychometric measure of health-related quality of life. Qual Life Res. 1999 May;8(3):209-24. doi: 10.1023/a:1008815005736. PMID 10472152
- [Background] Helms JE. An examination of the evidence in culturally adapted evidence-based or empirically supported interventions. Transcult Psychiatry. 2015 Apr;52(2):174-97. doi: 10.1177/1363461514563642. Epub 2014 Dec 22. PMID 25534401
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lara MA, Tiburcio M, Aguilar Abrego A, Sanchez-Solis A. A four-year experience with a Web-based self-help intervention for depressive symptoms in Mexico. Rev Panam Salud Publica. 2014 May-Jun;35(5-6):399-406. PMID 25211568
- [Background] Mira A, Breton-Lopez J, Garcia-Palacios A, Quero S, Banos RM, Botella C. An Internet-based program for depressive symptoms using human and automated support: a randomized controlled trial. Neuropsychiatr Dis Treat. 2017 Mar 31;13:987-1006. doi: 10.2147/NDT.S130994. eCollection 2017. PMID 28408833
- [Background] Munoz-Navarro R, Cano-Vindel A, Moriana JA, Medrano LA, Ruiz-Rodriguez P, Aguero-Gento L, Rodriguez-Enriquez M, Piza MR, Ramirez-Manent JI. Screening for generalized anxiety disorder in Spanish primary care centers with the GAD-7. Psychiatry Res. 2017 Oct;256:312-317. doi: 10.1016/j.psychres.2017.06.023. Epub 2017 Jun 12. PMID 28666201
- [Background] Osma J, Quilez-Orden A, Suso-Ribera C, Peris-Baquero O, Norman SB, Bentley KH, Sauer-Zavala S. Psychometric properties and validation of the Spanish versions of the overall anxiety and depression severity and impairment scales. J Affect Disord. 2019 Jun 1;252:9-18. doi: 10.1016/j.jad.2019.03.063. Epub 2019 Mar 29. PMID 30953927
- [Background] Parada F, Martinez V, Espinosa HD, Bauer S, Moessner M. Using Persuasive Systems Design Model to Evaluate "Cuida tu Animo": An Internet-Based Pilot Program for Prevention and Early Intervention of Adolescent Depression. Telemed J E Health. 2020 Feb;26(2):251-254. doi: 10.1089/tmj.2018.0272. Epub 2019 Jan 21. PMID 30668227
- [Background] Richards D, Timulak L, O'Brien E, Hayes C, Vigano N, Sharry J, Doherty G. A randomized controlled trial of an internet-delivered treatment: Its potential as a low-intensity community intervention for adults with symptoms of depression. Behav Res Ther. 2015 Dec;75:20-31. doi: 10.1016/j.brat.2015.10.005. Epub 2015 Oct 21. PMID 26523885
- [Background] Salamanca-Sanabria A, Richards D, Timulak L, Castro-Camacho L, Mojica-Perilla M, Parra-Villa Y. Assessing the efficacy of a culturally adapted cognitive behavioural internet-delivered treatment for depression: protocol for a randomised controlled trial. BMC Psychiatry. 2018 Feb 27;18(1):53. doi: 10.1186/s12888-018-1634-x. PMID 29482586
- [Background] Schroder J, Sautier L, Kriston L, Berger T, Meyer B, Spath C, Kother U, Nestoriuc Y, Klein JP, Moritz S. Development of a questionnaire measuring Attitudes towards Psychological Online Interventions-the APOI. J Affect Disord. 2015 Nov 15;187:136-41. doi: 10.1016/j.jad.2015.08.044. Epub 2015 Aug 28. PMID 26331687
- [Background] Tiburcio M, Lara MA, Aguilar Abrego A, Fernandez M, Martinez Velez N, Sanchez A. Web-Based Intervention to Reduce Substance Abuse and Depressive Symptoms in Mexico: Development and Usability Test. JMIR Ment Health. 2016 Sep 29;3(3):e47. doi: 10.2196/mental.6001. PMID 27687965
- [Background] Tiburcio M, Lara MA, Martinez N, Fernandez M, Aguilar A. Web-Based Intervention to Reduce Substance Abuse and Depression: A Three Arm Randomized Trial in Mexico. Subst Use Misuse. 2018 Nov 10;53(13):2220-2231. doi: 10.1080/10826084.2018.1467452. Epub 2018 May 16. PMID 29768070
- [Background] van Ballegooijen W, Cuijpers P, van Straten A, Karyotaki E, Andersson G, Smit JH, Riper H. Adherence to Internet-based and face-to-face cognitive behavioural therapy for depression: a meta-analysis. PLoS One. 2014 Jul 16;9(7):e100674. doi: 10.1371/journal.pone.0100674. eCollection 2014. PMID 25029507
- [Background] Wagner B, Horn AB, Maercker A. Internet-based versus face-to-face cognitive-behavioral intervention for depression: a randomized controlled non-inferiority trial. J Affect Disord. 2014 Jan;152-154:113-21. doi: 10.1016/j.jad.2013.06.032. Epub 2013 Jul 23. PMID 23886401
- [Background] Webb CA, Rosso IM, Rauch SL. Internet-Based Cognitive-Behavioral Therapy for Depression: Current Progress and Future Directions. Harv Rev Psychiatry. 2017 May/Jun;25(3):114-122. doi: 10.1097/HRP.0000000000000139. PMID 28475503
- [Background] mhGAP Intervention Guide for Mental, Neurological and Substance Use Disorders in Non-Specialized Health Settings: Mental Health Gap Action Programme (mhGAP): Version 2.0. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK390828/ PMID 27786430